CLINICAL TRIAL: NCT02934321
Title: Assessment of Satiety Following Oral Administration of an Erythritol Sweetened Beverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB201601141
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Satiety in Healthy Volunteers
Keywords: Erythritol; Satiety Response; Ghrelin
MeSH Terms: interventions — Erythritol; Aspartame

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspartame Sweetened Beverage (Active Comparator): Volunteers will consume a low-calorie, aspartame sweetened beverage (185 mg aspartame in water) after fasting for 10 hours and abstaining from alcohol, caffeine, and strenuous exercise for 24 hours prior to the visit.
  Interventions: Dietary Supplement: Aspartame
- Erythritol Sweetened Beverage (Experimental): Volunteers will consume an isosweet, compared to aspartame, high osmolar, low-calorie erythritol sweetened beverage (50.8 g erythritol in water, 1.66 Molar) after fasting for 10 hours and abstaining from alcohol, caffeine, and strenuous exercise for 24 hours prior to the visit.
  Interventions: Dietary Supplement: Erythritol

INTERVENTIONS:
Dietary Supplement: Erythritol — Erythritol is a well tolerated, low calorie sugar alcohol that is becoming more widely used as a sugar substitute.
  Arms: Erythritol Sweetened Beverage
Dietary Supplement: Aspartame — Aspartame is a well tolerated, commonly used artificial sweetener.
  Arms: Aspartame Sweetened Beverage

SUMMARY:
Erythritol is a low calorie sugar substitute that is being increasingly used to sweeten beverages and other food items. Greater amounts of erythritol are required to reach the sweetness level of a common soft drink as compared to aspartame, resulting in higher osmolarity for the erythritol sweetened beverage. Since associations have been noted between osmolarity and satiety, investigators propose that an erythritol sweetened beverage may enhance satiety more than a beverage sweetened with aspartame.

DETAILED DESCRIPTION:
The effects of an erythritol sweetened beverage on satiety has yet to be specifically explored. In this double-blind, 2-way crossover trial, healthy volunteers will consume one of two beverages on each visit: either an erythritol sweetened beverage or an aspartame sweetened beverage. Both beverages will be prepared to the same level of sweetness.

Timed blood samples will be collected over a period of two hours following consumption of the sweetened beverage. Serum total ghrelin and serum insulin will be measured from all blood samples. A validated hunger scale will be administered three times within the two hour period. Data analysis for all measures will be reported with respect to deviation from the initial baseline measured at time 0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI below 25
* Maintained a stable body weight for at least three months prior to volunteering

Exclusion Criteria:

* Exclude if smoking, substance abuse, have a chronic medical or psychiatric illness, regularly intake medications (except for oral contraceptives), regularly use supplements besides vitamins/minerals, have a history of gastrointestinal or renal disorders, have food allergies, have medical dietary restrictions, or have any abnormalities detected on physical examination indicative of disease.
* Participants must have intact gastrointestinal and kidney function to adequately absorb and eliminate the erythritol. Eligibility will be determined by self-reported medical history, physical examination, and specific questioning to exclude prior renal or Gastrointestinal disease after the informed consent process.
* Exclude if abnormal GI anatomy due to surgery (besides appendix removal) or congenital defect as may impair ghrelin production.
* Exclude if the patient is pregnant, lactating, or planning to become pregnant as erythritol has not been specifically tested in this population.
* Exclude if have a Body Mass Index over 25, as ghrelin as a marker of satiety may not be accurate at high Body Mass Index.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Ghrelin taken over 2 hours post beverage total area under curve (AUC) | 0 min, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 60 min, 75 min, 90 min, 120 min following consumption of test drink

SECONDARY OUTCOMES:
Ghrelin minimum concentration | 0 min, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 60 min, 75 min, 90 min, 120 min following consumption of test drink
Serum insulin concentration | 0 min, 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 60 min, 75 min, 90 min, 120 min following consumption of test drink
Change in hunger rating scale | 0 min, 30 min, 120 min following consumption of test drink

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Brantly, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Clinical Research Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No